CLINICAL TRIAL: NCT07299123
Title: Efficacy and Safety of Sequential Infusion of Hypoxic 3D-Cultured Umbilical Cord Mesenchymal Stem Cells in Haploidentical Hematopoietic Stem Cell Transplantation for Severe Aplastic Anemia: A Multicenter, Randomized, Phase 1 Trial
Brief Title: Phase I Clinical Study of Haplo-HSCT Combined With Hypoxic 3D-Cultured Umbilical Cord MSC for the Treatment of SAA
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: The Fourth Medical Center of Chinese PLA General Hospital (Unknown); Beijing 302 Hospital (Other); The First Medical Center of Chinese PLA General Hospital (Other); Pollon Life Co., Ltd. (Unknown); Yan'an University Affiliated Hospital (Other); The University of Hong Kong-Shenzhen Hospital (Other); Beijing Friendship Hospital (Other); Beijing GeniusCure Biotechnology Co., Ltd. (Unknown); Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, Jian Bo, Chief Physician / Associate Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S2021-384-01
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Severe Aplastic Anemia (SAA); Severe Aplastic Anemia, Refractory; Severe Aplastic Anemia
Keywords: Severe Aplastic Anemia; Hematopoietic Stem Cell Transplantation; Mesenchymal Stem Cells
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D hypoxia-preconditioned UC-MSC group (Experimental)
  Interventions: Drug: 3D hypoxia-preconditioned UC-MSC group
- 2D UC-MSC group (Active Comparator)
  Interventions: Drug: 2D UC-MSC group

INTERVENTIONS:
Drug: 3D hypoxia-preconditioned UC-MSC group — 5 × 10⁵/kg 3D hypoxia-preconditioned UC-MSCs at 4 h before HSC infusion
  Arms: 3D hypoxia-preconditioned UC-MSC group
Drug: 2D UC-MSC group — 5 × 10⁵/kg 2D UC-MSCs at 4 h before HSC infusion
  Arms: 2D UC-MSC group

SUMMARY:
Efficacy and Safety of Sequential Infusion of Hypoxic 3D-Cultured Umbilical Cord Mesenchymal Stem Cells in Haploidentical Hematopoietic Stem Cell Transplantation for Severe Aplastic Anemia: A Multicenter, Randomized, Phase 1 Trial

DETAILED DESCRIPTION:
The enrolled patients with an HLA-haploidentical relative for HSCT received the fludarabine (Flu) + cyclophosphamide (Cy) + antithymocyte globulin (ATG) conditioning regimen. For the patients with acute SAA (SAA-I), intravenous administration of 30 mg/(m2 day) of Flu and 500-800 mg/(m2 day) of Cy was performed from days -5 to -2, and 5μg/(kg day) of ATG was administered from days -4 to -1. For the patients with chronic SAA (SAA-II), the same treatment of ATG and Cy was applied as above with the supplement of 0.6 mg/(kg 6 h) of busulfan (BU) from days -8 to -5 prior to transplantation. Donor selection and hematopoietic stem cell mobilization and collection were conducted based on the consensus of The Chinese Society of Hematology regarding indications, conditioning regimens, and donor selection for allogeneic hematopoietic stem cell transplantation. On day 0, HSCs were infused intravenously. Both groups received 5 × 10⁵/kg UC-MSCs at 4 h before HSC infusion. The control group was transfused with conventional 2D-cultured UC-MSCs, whereas the experimental group received 3D hypoxia-preconditioned UC-MSCs. Standard GVHD prophylaxis consisted of mycophenolate mofetil, cyclosporine A, and methotrexate (MTX).

ELIGIBILITY:
The inclusion criteria were (1) age 6 to 60 years; (2) diagnosis of SAA or very SAA according to the International Aplastic Anemia Study Group[21]; (3) without any severe pulmonary, cardiac, liver, or renal diseases or any active infection; and (4) adequate performance status (Eastern Cooperative Oncology Group score 0-2). Exclusion Criteria：(1)Age 6 years or > 60 years; (2)Failure to meet the IAASG-defined diagnosis of SAA/vSAA, or confirmed (3)Fanconi anemia, congenital aplastic anemia (e.g., dyskeratosis congenita, Diamond-Blackfan anemia); (4)Presence of severe pulmonary, cardiac, hepatic, or renal insufficiency; Uncontrolled active infection; (5)Eastern Cooperative Oncology Group (ECOG) performance status score ≥ 3.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | The incidence and severity of adverse events (AEs) within the first 150 days after haplo-HSCT

SECONDARY OUTCOMES:
acute GVHD | 100days after HSCT
chronic GVHD | 1 years after HSCT
Surivial | 1 year after HSCT
Rates of relapse | UP to 2 years after HSCT
The implantation | Up to 4 weeks after HSCT
  The implantation rate and implantation time.

CONTACTS AND LOCATIONS:
Locations (1):
- 28 Fuxing Road, Beijing, China., Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Treatment effect
Supporting Information: Study Protocol
Time Frame: 2025/10/1-2027/1/1

DOCUMENTS (1):
  • Study Protocol (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT07299123/Prot_000.pdf